CLINICAL TRIAL: NCT05337319
Title: A Multi-center, Prospective, Registry Study to Estimate the Current Status of Care for Patients With Coronary Artery Disease
Brief Title: Prospective Registry of the Current Status of Care for Patients With Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Principal Investigator, Beijing Anzhen Hospital
Other Study IDs: NCCMRC202201_001
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will estimate the current status of care for participants with coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with discharge diagnosis as coronary artery disease (including atherosclerosis or non-athrosclerosis)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The overall composite of 10 performance measures for CAD care | Duration of hospital stay, an expected average of 1 week
  Performance measures for CAD care including:
  Proportion of patients received fibrinolytic therapy within 30 mins (STEMI) Proportion of patients received primary percutaneous coronary intervention within 90 mins (STEMI) Proportion of patients received reperfusion therapy (STEMI, high or moderate risk NSTE-ACS) Proportion of patients with aspirin prescribed at discharge Proportion of patients with P2Y12 inhibitors prescribed at discharge Proportion of patients with beta-blocker prescribed at discharge Proportion of patients with statin prescribed at discharge Proportion of left ventricular systolic dysfunction patients with ACEI or ARB prescribed at discharge Proportion of patients received evaluation of left ventricular systolic function Proportion of patients with a diagnosed non-obstructive coronary artery disease at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Shaoping Nie, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China